CLINICAL TRIAL: NCT03109275
Title: Connectome Characterization With Aging Using Functional and Structural MRI
Brief Title: Connectome Characterization With Aging
Acronym: AGE-CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0687
Record Dates: First submitted 2017-03-01; First posted 2017-04-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single MRI examination (Active Comparator): 40 subjects will benefit from a full MRI
  Interventions: Other: Single complete MRI intervention
- Reproducibility study (Sham Comparator): 10 subjects will benefit from the realization of 3 MRI. An MRI examination performed at the time of inclusion and then an examination, at 3 months and at 9 months (ie 3 examinations per subject).
  Interventions: Other: Single complete MRI intervention

INTERVENTIONS:
Other: Single complete MRI intervention — MRI examination will comprise conventional T1 and FLAIR sequences, and advanced sequences such as rs-fMRI and High angular resolution MRI (HARDI).

SUMMARY:
The main aim of this project is to develop a new model to characterize brain connectivity and its changes with aging. This characterization will be based on new sensitive and specific markers, allowing a better understanding of structural and functional brain networks. To this end, two complementary MRI methods will be developed: 1) Resting-state functional MRI (rs-fMRI) which allows the measurement of cerebral activity in different cortical gray matter regions, and 2) high angular resolution diffusion imaging (HARDI) MRI, which allows to characterize brain tissue microarchitecture. HARDI sequences will be developed to acquire and reconstruct fiber tractography of patient's brains. In combination with conventional MRI, both HARDI and rs-fMRI will be used to estimate the connection degree between each pair of cortical regions, so- called "Connectome". Once generated, brain networks will be quantified through numerous graph metrics, such as graph density, global efficiency and assortativity (etc.), reflecting the organization and topology of subjects' connectivity with aging.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers (Men and women) aged between 18 and 50 years
* No neurological or psychiatric diseases

Exclusion Criteria:

* MRI contraindications
* Pregnant women or nursing women
* Persons under guardianship or any other administrative or deprivation of liberty or of right

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Functional and structural connectivity MRI marker : resting-state fMRI | End of study (one year)
  Functional connectivity of grey matter (GM) using resting-state fMRI
Functional and structural connectivity MRI marker : Functional connectivity | End of study (one year)
  Graph-theory methods analysis of functional connectivity of grey matter
Functional and structural connectivity MRI marker : Diffusion tensor | End of study (one year)
  Structural connectivity of white matter (WM) fiber bundles measured by diffusion tensor imaging
Functional and structural connectivity MRI marker : Structural connectivity | End of study (one year)
  Graph-theory methods analysis of Structural connectivity of white matter (WM) fiber
Functional and structural connectivity MRI marker : SPM software | End of study (one year)
  Cortical and subcortical grey matter (GM) volumes using the SPM software

SECONDARY OUTCOMES:
Metrics of functional connectivity | End of study (one year)
  Calculation of functional connectivity metrics using graphs theory methods

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mouchet-Mages, MD, Principal Investigator — CH le Vinatier
Locations (1):
- CH le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nusbaum F, Hannoun S, Barile B, Suprano I, Mouchet S, Sappey-Marinier D. Personal Income Performance Correlates with Brain Structural Network Modularity but Not Intelligence Quotient. Brain Connect. 2024 Jun;14(5):284-293. doi: 10.1089/brain.2023.0077. Epub 2024 Jun 7. PMID 38848246